CLINICAL TRIAL: NCT04457895
Title: A Randomized, Open-labelled, Controlled Trial Evaluating the Efficacy of a Physical Therapy-yoga-patient Educational Program for Breast Cancer Patients With Pain Due to Hormonal Therapy Treatment.
Brief Title: Evaluation of the Efficacy of a Physical Therapy-yoga-patient Educational Program for Breast Cancer Patients With Pain Due to Hormonal Therapy Treatment.
Acronym: SKYPE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2020-05 SKY
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; hormonotherapy; osteo articular pain; yoga; patient educational project
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): For experimental arm patients, there will be a 90-min yoga-therapeutic education session/week (during 6 weeks) given by a physical therapist trained to postural yoga (the first on site and by videoconference for the others).
  Starting the first day of the yoga practice there will be one daily 15 min session at home with "My Yoga Guide" and the audio guide during 12 weeks.
  Interventions: Behavioral: educational yoga program
- control arm (Placebo Comparator): The control arm patients will have standard care. They will be proposed to participate in the physical therapy - yoga - educational program after the end of the study.
  Interventions: Other: no intervention

INTERVENTIONS:
Behavioral: educational yoga program — Daily 15-min yoga sessions at home with the "Le guide du yoga" and the audio-guide, during 12 weeks.
  One 90-min yoga-therapeutic education session/week (during 6 weeks) given by a physical therapist trained to postural yog (the first on site and by videoconference for the others)
  Arms: Experimental arm
Other: no intervention — no yoga session at home and no yoga -therapeutic educatuion session
  Arms: control arm

SUMMARY:
As much as 50% of patients treated with hormonotherapy (HT) for breast cancer (BC) suffer from osteoarticular pain during treatment. Secondary effects have become a real issue because of their consequences on the patients' quality of life, but also on treatment efficacy and survival when they induce dose reduction or premature withdrawal of treatment.

Additional medicines (acupuncture, hypnosis, yoga) have become more and more popular these last years. 48 to 80% of patients with BC eventually choose them. A review comparing efficacy of various therapies to decrease osteoarticular pain concludes to a highest efficacy of anti-inflammatory treatments, paracetamol and yoga.

It thus appears innovative to complete this care with a patient educational project (PEP) in postural yoga instructed by a trained physical therapist, which will enable patients to practice yoga postures at home by themselves.

The investigators conducted a pilot study "SKYPE" with 24 algic patients treated with HT after BC, whose results are very promising.

The investigators now propose in the continuity of the pilot study a multicenter randomized controlled study comparing the efficacy of SKYPE care on pain reduction, an educative care combining physical therapy and yoga, to a control group in patients treated with HT for a BC with osteoarticular and/or musculoskeletal pain.

Furthermore, in order to examine whether yoga interventions may influence inflammation through their effects on the level of a wide range of pro- and anti-inflammatory cytokines (30), the investigators will Change in circulating cytokines' level between baseline level (T0) and post-treatment level (T2) in both groups will be analyzed and if so correlation will be established.

DETAILED DESCRIPTION:
Numerous initiatives have started in France, often associative. It is essential to evaluate in a rigorous manner, these therapies before making them part of the patient's care pathway.

Yoga has shown a real benefit in terms of pain reduction in patients with BC treated with HT. These osteoarticular pains are the secondary effect on which a physical therapeutic care can have a real benefit.

It thus appears innovative to complete this care with a therapeutic education program (TEP) in postural yoga which will enable patients to practice yoga postures at home by themselves. Yoga allows a large adaptation to pains expressed by each patient. It will favor the development of the feeling of control that they have in particular on their pain. participants will so improve the self-efficacy, the quality of life, and will reduce their fatigue and their pain. The patients involved have already lived major body transformations because of the disease and treatments. Yoga will help them put their lives together again, both physically and psychologically, and reclaim their body.

Studies have shown the short-term effects of yoga practice on anxiety, stress, pain and quality of life. Few rare studies have suggested that patients could add yoga practice at home to the supervised sessions, but these studies lacked therapeutic patient education. To date, to our knowledge, no data on the effect of the realization of yoga postures at home on increase of the patients' self-competency feeling are available in France. Also, the long-term effects of such programs need to be assessed.

The Montpellier Cancer Institute (ICM) has set-up 8 years ago yoga sessions for women with breast cancer, together with an association located in Montpellier.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non metastatic breast cancer
* Ongoing hormone therapy, with no treatment modification in the 30 days before inclusion
* Osteoarticular and/or musculoskeletal pain due to HT ≥ 4 on the Numeric Pain Rating Scale (NPRS)
* Previous treatment (surgery, chemotherapy or radiotherapy) ended at least 2 months before inclusion
* Informed patient and signed informed consent received
* Affiliation to a social security system

Exclusion Criteria:

* Chronic rhumatologic pain with specific care needed
* Regular Yoga practice in the 3 months before inclusion
* Contraindication or clinical state not allowing physical practice
* Patient whose regular follow-up is initially impossible for psychological, family, social or geographical reasons,
* Pregnant and breastfeeding woman

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
the efficacy of a combined intervention of physical therapy and yoga, including patient education with a control group for confirmed osteoarticular and/or musculoskeletal pain (≥4) due to hormone therapy in patients treated for breast cancer. | 12 weeks
  Rate of patients with a 2-point reduction on the Numeric Pain Rating Scale (NPRS) of osteoarticular and/or musculoskeletal pain due to hormonal therapy treatment between T0 (inclusion) and T2 (end of treatment).

SECONDARY OUTCOMES:
the evolution of osteoarticular and/or musculoskeletal pain characteristics related to hormone therapy | 12 weeks
  The evolution of osteoarticular and/or musculoskeletal pain characteristics will be described according to the questionnaire "BPI- Brief Pain Inventory"
the patient compliance at yoga-therapeutic education session and yoga self-practice | 12 weeks
  The patient attendance at yoga-therapeutic education session and yoga self-practice will be noted on the logbooks filled out by the patients.
the reasons for adhesion or non-adhesion to yoga self-practice | 12 weeks
  The reasons why patients practice or do not practice yoga at home will be noted on the logbooks filled out by the patient
To assess forward-flexion flexibility | 12 weeks
  Forward-flexion flexibility is defined by the distance between the fingertips and the floor. It will be measured with a ruler.
To assess respiratory capacity | 12 weeks
  Respiratory capacity will be measured with a spirometer (Forced Expiratory Volume in 1 second (FEV1)
the hormone therapy treatment and its compliance | 12 weeks
  Taking hormonotherapy treatments will be reported in a log-book by the patients
to assess quality of life by short form questionnaire | 12 weeks
  Quality of life will be measured by EORTC SF-36 questionnaire (European Organisation for Research and Treatment of Cancer, Short Form)
to assess quality of life by Quality of Life Questionnaire | 12 weeks
  Quality of life will be measured by EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire)
to assess quality of life by Quality of Life Questionnaire specify for Breast Cance | 12 weeks
  Quality of life will be measured by EORTC QLQ-BR23 questionnaires (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire specify for Breast Cancer)
to assess fatigue | 12 weeks
  Fatigue will be measured by the Fatigue dimension of the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire) questionnaire
anxiety and depression | 12 weeks
  Anxiety and depression will be measured by HADS scale (Hospital Anxiety and Depression Scale) (if score or = 9, result is no significant, if sore is between 10 and 12, result is limit, if result is > or = 13, result is significant)
the induced self-competence feeling | 12 weeks
  The self-competence feeling induced will be assessed using the GSES (General Self Efficacy-Schwarzer) questionnaire (10 questions - scale 1- not at all true to 4-totally true)
the patients' satisfaction towards the program | 12 weeks
  Satisfaction will be measured using the Likert scale (0 no satisfy to 10: strongly satisfy
the patient's inflammatory biological profile | 12 weeks
  The inflammatory biological profile of the patient will be determined by correlation of cytokine levels at the beginning (T0) and end (T2) of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Faravel, Study Chair — ICM Val d'Aurelle
Locations (7):
- France (7):
  - CH Libourne, Libourne, Aquitaine
  - Icm Val D'Aurelle, Montpellier, Herault
  - CHU Nîmes, Nîmes, Herault
  - Insitut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle,
  - Institut Bergonié, Bordeaux, Nouvelle-Aquitaine
  - Institut du sein Basque, Tosse, Nouvelle-Aquitaine
  - Institut de Cancérologie de l'Ouest, Angers, Pays de la Loire Region

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after coding by an inclusion number, 1st letter of the surname and first name can be shared.
  Participant data will be available upon request and with the completion of a contract between the sponsor and the applicant.
  The study protocol, the statistical analysis plan and the analytical code may also be subject to data sharing under a transfer contract (EU-MCR).

REFERENCES:
- [Background] Lintermans A, Van Asten K, Wildiers H, Laenen A, Paridaens R, Weltens C, Verhaeghe J, Vanderschueren D, Smeets A, Van Limbergen E, Leunen K, Christiaens MR, Neven P. A prospective assessment of musculoskeletal toxicity and loss of grip strength in breast cancer patients receiving adjuvant aromatase inhibitors and tamoxifen, and relation with BMI. Breast Cancer Res Treat. 2014 Jul;146(1):109-16. doi: 10.1007/s10549-014-2986-7. Epub 2014 May 11. PMID 24816806
- [Background] Peppone LJ, Janelsins MC, Kamen C, Mohile SG, Sprod LK, Gewandter JS, Kirshner JJ, Gaur R, Ruzich J, Esparaz BT, Mustian KM. The effect of YOCAS(c)(R) yoga for musculoskeletal symptoms among breast cancer survivors on hormonal therapy. Breast Cancer Res Treat. 2015 Apr;150(3):597-604. doi: 10.1007/s10549-015-3351-1. Epub 2015 Mar 27. PMID 25814054
- [Background] Crew KD, Greenlee H, Capodice J, Raptis G, Brafman L, Fuentes D, Sierra A, Hershman DL. Prevalence of joint symptoms in postmenopausal women taking aromatase inhibitors for early-stage breast cancer. J Clin Oncol. 2007 Sep 1;25(25):3877-83. doi: 10.1200/JCO.2007.10.7573. PMID 17761973
- [Background] Lyman GH, Greenlee H, Bohlke K, Bao T, DeMichele AM, Deng GE, Fouladbakhsh JM, Gil B, Hershman DL, Mansfield S, Mussallem DM, Mustian KM, Price E, Rafte S, Cohen L. Integrative Therapies During and After Breast Cancer Treatment: ASCO Endorsement of the SIO Clinical Practice Guideline. J Clin Oncol. 2018 Sep 1;36(25):2647-2655. doi: 10.1200/JCO.2018.79.2721. Epub 2018 Jun 11. PMID 29889605
- [Background] Lombard JM, Zdenkowski N, Wells K, Beckmore C, Reaby L, Forbes JF, Chirgwin J. Aromatase inhibitor induced musculoskeletal syndrome: a significant problem with limited treatment options. Support Care Cancer. 2016 May;24(5):2139-2146. doi: 10.1007/s00520-015-3001-5. Epub 2015 Nov 10. PMID 26556210
- [Background] Galantino ML, Desai K, Greene L, Demichele A, Stricker CT, Mao JJ. Impact of yoga on functional outcomes in breast cancer survivors with aromatase inhibitor-associated arthralgias. Integr Cancer Ther. 2012 Dec;11(4):313-20. doi: 10.1177/1534735411413270. Epub 2011 Jul 6. PMID 21733988
- [Background] Sharma M, Lingam VC, Nahar VK. A systematic review of yoga interventions as integrative treatment in breast cancer. J Cancer Res Clin Oncol. 2016 Dec;142(12):2523-2540. doi: 10.1007/s00432-016-2269-2. Epub 2016 Sep 15. PMID 27630024
- [Background] Cramer H, Lauche R, Klose P, Lange S, Langhorst J, Dobos GJ. Yoga for improving health-related quality of life, mental health and cancer-related symptoms in women diagnosed with breast cancer. Cochrane Database Syst Rev. 2017 Jan 3;1(1):CD010802. doi: 10.1002/14651858.CD010802.pub2. PMID 28045199
- [Background] Kiecolt-Glaser JK, Bennett JM, Andridge R, Peng J, Shapiro CL, Malarkey WB, Emery CF, Layman R, Mrozek EE, Glaser R. Yoga's impact on inflammation, mood, and fatigue in breast cancer survivors: a randomized controlled trial. J Clin Oncol. 2014 Apr 1;32(10):1040-9. doi: 10.1200/JCO.2013.51.8860. Epub 2014 Jan 27. PMID 24470004
- [Background] Chandwani KD, Perkins G, Nagendra HR, Raghuram NV, Spelman A, Nagarathna R, Johnson K, Fortier A, Arun B, Wei Q, Kirschbaum C, Haddad R, Morris GS, Scheetz J, Chaoul A, Cohen L. Randomized, controlled trial of yoga in women with breast cancer undergoing radiotherapy. J Clin Oncol. 2014 Apr 1;32(10):1058-65. doi: 10.1200/JCO.2012.48.2752. Epub 2014 Mar 3. PMID 24590636
- [Background] Greenlee H, Balneaves LG, Carlson LE, Cohen M, Deng G, Hershman D, Mumber M, Perlmutter J, Seely D, Sen A, Zick SM, Tripathy D; Society for Integrative Oncology. Clinical practice guidelines on the use of integrative therapies as supportive care in patients treated for breast cancer. J Natl Cancer Inst Monogr. 2014 Nov;2014(50):346-58. doi: 10.1093/jncimonographs/lgu041. PMID 25749602
- [Background] Olsson Moller U, Beck I, Ryden L, Malmstrom M. A comprehensive approach to rehabilitation interventions following breast cancer treatment - a systematic review of systematic reviews. BMC Cancer. 2019 May 20;19(1):472. doi: 10.1186/s12885-019-5648-7. PMID 31109309
- [Background] Felson DT, Cummings SR. Aromatase inhibitors and the syndrome of arthralgias with estrogen deprivation. Arthritis Rheum. 2005 Sep;52(9):2594-8. doi: 10.1002/art.21364. No abstract available. PMID 16142740
- [Background] Bower JE, Irwin MR. Mind-body therapies and control of inflammatory biology: A descriptive review. Brain Behav Immun. 2016 Jan;51:1-11. doi: 10.1016/j.bbi.2015.06.012. Epub 2015 Jun 23. PMID 26116436
- [Background] Djalilova DM, Schulz PS, Berger AM, Case AJ, Kupzyk KA, Ross AC. Impact of Yoga on Inflammatory Biomarkers: A Systematic Review. Biol Res Nurs. 2019 Mar;21(2):198-209. doi: 10.1177/1099800418820162. Epub 2018 Dec 20. PMID 30572710
- [Background] Bower JE, Greendale G, Crosswell AD, Garet D, Sternlieb B, Ganz PA, Irwin MR, Olmstead R, Arevalo J, Cole SW. Yoga reduces inflammatory signaling in fatigued breast cancer survivors: a randomized controlled trial. Psychoneuroendocrinology. 2014 May;43:20-9. doi: 10.1016/j.psyneuen.2014.01.019. Epub 2014 Jan 30. PMID 24703167
- [Background] Long Parma D, Hughes DC, Ghosh S, Li R, Trevino-Whitaker RA, Ogden SM, Ramirez AG. Effects of six months of Yoga on inflammatory serum markers prognostic of recurrence risk in breast cancer survivors. Springerplus. 2015 Mar 26;4:143. doi: 10.1186/s40064-015-0912-z. eCollection 2015. PMID 25853030
- [Background] Rao RM, Vadiraja HS, Nagaratna R, Gopinath KS, Patil S, Diwakar RB, Shahsidhara HP, Ajaikumar BS, Nagendra HR. Effect of Yoga on Sleep Quality and Neuroendocrine Immune Response in Metastatic Breast Cancer Patients. Indian J Palliat Care. 2017 Jul-Sep;23(3):253-260. doi: 10.4103/IJPC.IJPC_102_17. PMID 28827927
- [Background] Faravel K, Jarlier M, Meignant L, Thomaso M, Del Rio M, Jacot W, Stoebner A. Efficacy of a physiotherapy, yoga and patient education programme for patients with breast cancer and hormone therapy-induced pain: a multicentre randomised study protocol (SKYPE 2). BMJ Open. 2024 Jan 8;14(1):e075378. doi: 10.1136/bmjopen-2023-075378. PMID 38191246
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669